CLINICAL TRIAL: NCT06192771
Title: Feasibility of Early Swallowing and Speech Intervention for Head and Neck Cancer Patients Treated SURGically
Acronym: ESSI-SURG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Rosemary Martino, PhD, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-5503
Record Dates: First submitted 2023-12-05; First posted 2024-01-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: Dysphagia; Head and Neck Cancer
Keywords: dysphagia; head and neck cancer; speech language pathology; surgery; speech; early intervention; medical outcomes
MeSH Terms: conditions — Deglutition Disorders; Head and Neck Neoplasms; Speech | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Control (Active Comparator): Participants in this Arm will receive the current standard of care, which includes a referral to SLP in response to suspicion of a swallowing problem from either assessment by the medical team and/or patient report.
  Interventions: Behavioral: Standard-of-Care
- Arm 2 - Intervention (Experimental): Participants in this Arm will receive the ESSI-SURG behavioural intervention by a live SLP.
  Interventions: Behavioral: ESSI-SURG

INTERVENTIONS:
Behavioral: ESSI-SURG — Patients will receive 3 face-to-face sessions with a speech-language pathologist (SLP), each with a specific goal, namely: pre-surgical educational, a post-operative day 3 therapy, and post-operative day 7 therapy. Following discharge from hospital, participants will be seen by an SLP for 4 weekly sessions, offered via telehealth or face-to-face depending on the patient's clinic schedule and/or availability.
  Arms: Arm 2 - Intervention
Behavioral: Standard-of-Care — Participants will receive the current standard of care, which includes a referral to SLP in response to suspicion of a swallowing problem from either assessment by the medical team and/or patient report.
  Arms: Arm 1 - Control

SUMMARY:
Oral cavity cancer (OCC) is one of the most common cancers worldwide, with tongue cancer being one of the most common subtypes. Patients with oral cancers can experience painful swallowing, swallowing difficulty (dysphagia), and associated weight loss long after surgery. Not only is dysphagia an independent predictor of quality of life (QoL) in cancer survivorship, it can also have a devastating impact on the health of patients resulting from complications such as pneumonia, malnutrition and feeding tube dependence. Emerging evidence suggests that patients undergoing surgery benefit from engaging with speech-language pathologists (SLPs) before problems arise, to learn swallow strategies that may become useful in their rehabilitation. This in turn has the potential to reduce complications and minimize the length of feeding tube dependency.

This study will assess the feasibility of conducting a prospective clinical trial that would evaluate the effects on patient health, function and overall benefit of early and systematic SLP speech and swallowing intervention for head and neck cancer patients planned for curative surgical treatment. We will also assess long-term changes in select clinical and patient-reported outcomes comparing their status before, and one month after, treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with at least T2 stage tongue SCC who are planned for partial glossectomy and free flap reconstruction and are anticipated to achieve a post-operative independent oral intake.
* Proficient in spoken and written English

Exclusion Criteria:

* Patients who are planned for total glossectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Study feasibility as measured by rate of accrual | Baseline to Post-Discharge Week 5
  Feasibility success will be defined as the following across all patients and compared by arm: an accrual rate >90%.
Study feasibility as measured by attrition | Baseline to Post-Discharge Week 5
  Feasibility success will be defined as the following across all patients and compared by arm: an attrition rate of <10%.
Study feasibility as measured by data fidelity for clinician assessments | Baseline to Post-Discharge Week 5
  Feasibility success will be defined as the following across all patients and compared by arm: data fidelity rate of >80% for clinical assessments.
Study feasibility as measured by data fidelity for patient-reported outcomes | Baseline to Post-Discharge Week 5
  Feasibility success will be defined as the following across all patients and compared by arm: data fidelity rate of >90% for patient reported outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Martino, PhD, Principal Investigator — University Health Network, Toronto; Jonathan Irish, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada